CLINICAL TRIAL: NCT06468319
Title: Assessment of Pregnancy Outcomes Through Demographic Surveillance and Prospective Data Collection at a Health Facility in Kalifabougou, Mali
Brief Title: Pregnancy Registry in Mali
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/84/CE/USTTB
Record Dates: First submitted 2024-05-28; First posted 2024-06-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Malaria; Pregnancy Related
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood collection for baseline hemoglobin and malaria infection status. Urine and/or serum collection for pregnancy test. Collection of placenta for malaria testing and pathology/histology. Cord blood collection for malaria infection status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Community Census Cohort: Women of child-bearing aged (WOCBA) identified within the community.
- Health Facility Cohort: Pregnant women presenting at the health facility for antenatal care or referred in from the Community Consensus Cohort.
- Offspring from Health Facility Cohort: Children born to women in the health facility cohort.

SUMMARY:
This registry will assess pregnancy outcomes through demographic surveillance and prospective data collection at a health facility in Kalifabougou, Mali.

DETAILED DESCRIPTION:
This pregnancy registry will gather background data on pregnancy rates and outcomes as well as infant health data to inform future implementation of clinical trials testing monoclonal antibodies (mAbs) to prevent malaria in pregnancy.

In the first part of the study (Community Census Cohort), women of child-bearing age (WOCBA) in the community will be identified and followed for up to 3 years to detect pregnancy at all stages. Upon detection of pregnancy, these women may then transition to participation in the Health Facility Cohort.

In the second part of the study (Health Facility Cohort), data will be prospectively collected from pregnant women presenting at the health facility for antenatal care (ANC) visits or referred in from the Community Census Cohort. The pregnant women will be followed through pregnancy outcome and until 12 months postpartum, and their infant(s) will be followed until 12 months of age.

The study team will collect baseline information in a systematic manner on early pregnancy events, pregnancy and postpartum complications and outcomes, utilization of existing malaria prevention tools, malaria infections and clinical disease, birth outcomes, and follow-up of subsequent offspring.

ELIGIBILITY:
Inclusion Criteria:

Community Census Cohort:

1. Females of childbearing potential or pregnant females.
2. Aged 15 to 49 years.
3. Able to provide verbal individual informed consent.

Health Facility Cohort:

1. Pregnant females 15 to 49 years and their subsequent offspring.
2. Resides in or in the health catchment area of Kalifabougou and willing to return to the health center for Antenatal Care (ANC) visits.
3. Able to provide written individual informed consent for herself and her future offspring(s).

Exclusion Criteria:

Community Census Cohort:

1. Temporary residence in the study area.
2. Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of an individual participating in the study, interfere with the evaluation of the study objectives, or render the participant unable to comply with the protocol.

Health Facility Cohort:

1. Temporary residence in the study area.
2. Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of an individual participating in the study, interfere with the evaluation of the study objectives, or render the participant unable to comply with the protocol.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Malian females of childbearing age (15-49 years) Community Census Cohort: 4000 unique women Health Facility Cohort: 2500 unique women (inclusive of women who transition for enrollment from the Community Census Cohort)
  Offspring from Health Facility Cohort: 3000 children
Sampling Method: Non-Probability Sample
Enrollment: 9500 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Number of pregnancies | Through study completion, an average of 1 year
  Detected by urine or serum by active and passive screening
Number of malaria cases | Through study completion, an average of 1 year
  Detected by RDT and/or blood smear and/or PCR during pregnancy defined as any parasitemia with or without malaria symptoms
Incidence of placental malaria | Through study completion, an average of 1 year
  Detected by blood smear or pathology/histology, at delivery
Use of other malaria prevention tools | Through study completion, an average of 1 year
  Recorded by survey
Number of Participants with anemia during pregnancy and post-partum | Through study completion, an average of 1 year
  Defined as hemoglobin level less than 11 g/dL
Dating of pregnancies | Through study completion, an average of 1 year
  Measured at each ANC visit by ultrasound and last menstrual period
Number of Maternal Deaths | Through study completion, an average of 1 year
Number of fetal Losses and Stillbirths | Through study completion, an average of 1 year
  Pregnancies terminated in the first trimester (<=12 weeks) and in the second trimester (>12 and <28 weeks) and stillbirth
Number of multiple gestations | Through study completion, an average of 1 year
  Twins, triplets, or multiple gestations during pregnancy
Incidence of preterm delivery | Through study completion, an average of 1 year
  Preterm delivery (≥28 to <37 weeks)
Occurrence of chronic medical conditions | Through study completion, an average of 1 year
  Description and reporting of occurrence of chronic medical conditions during pregnancy and/or post-partum
Occurrence of pregnancy and post-partum adverse outcomes | Through study completion, an average of 1 year
  Description and reporting of occurrence of pregnancy and post-partum adverse outcomes including but not limited to gestational diabetes, gestational hypertension, pre-eclampsia, eclampsia, postpartum hemorrhage, and postpartum depression

SECONDARY OUTCOMES:
Number of neonatal deaths | Through study completion, an average of 1 year
  Neonatal death as defined as early (≤7 days) or late (>7 days ≤28 days) after delivery
Incidence of low Birth Weight (LBW) | Through study completion, an average of 1 year
  LBW as defined as <2.5 kg at birth
Incidence of preterm birth | Through study completion, an average of 1 year
  Preterm birth (≥28 to <37 weeks)
Occurrence and description of malformations | Through study completion, an average of 1 year
  Occurrence and description of malformations identified at delivery and within the first 6 months of life
Occurrence of Small for Gestational Age (SGA) | Through study completion, an average of 1 year
  defined as newborns whose birth weight is <10th percentile for gestational age as defined by INTERGROWTH-21st international standards
Occurrence of malaria (symptomatic and asymptomatic) in neonates and infants | Through study completion, an average of 1 year
  Detected by RDT and/or blood smear and/or PCR at birth and throughout first year of life defined as any parasitemia with or without malaria symptoms
Occurrence of anemia during infancy at 6 and 12 months of age | Through study completion, an average of 1 year
  Anemia during infancy as defined by age of testing
Occurrence of neonatal/infant/pediatric adverse outcomes | Through study completion, an average of 1 year
  Description and reporting of occurrence of neonatal/infant/pediatric adverse outcomes
Timing of receipt of routine vaccinations | Through study completion, an average of 1 year
  Reporting and timing of receipt of routine vaccinations, including malaria vaccines, and other standard of care anti-malarial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kassoum Kayentao, MD, MPH, PhD, Principal Investigator — Faculté de Médecine Pharmacie d'Odontostomatologie (FMOS); Peter Crompton, MD, MPH, Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- Kalifabougou MRTC Clinic, Kalifabougou, Koulikoro, Mali

IPD SHARING:
Plan to Share IPD: Undecided